CLINICAL TRIAL: NCT02767609
Title: Measuring Cerebral Blood Flow Using Pseudo-continuous Arterial Spin Labeling Perfusion Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Brenda Bartnik Olson, PhD, Associate Proffesor, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5140083
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Traumatic Brain Injury; Multiple Sclerosis; Alzheimer's Disease; Tumor
MeSH Terms: conditions — Brain Injuries, Traumatic; Multiple Sclerosis; Alzheimer Disease; Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magentic Resonance Imaging (Experimental): magnetic Resonance Imaging.
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — All participants will have be given a MRI using a pseudo-continuous arterial spin labeling perfusion sequence.

SUMMARY:
This study will test a new MRI sequence that measures cerebral blood flow (CBF). Because this technique for measuring CBF is new, there is little information on what the normal values for different regions of the brain should be. Information from the study will be used to establish normative CBF values for the brain, improving the reliable use of this technique for the diagnosis of brain injury or disease.

DETAILED DESCRIPTION:
Cerebral blood flow (CBF) represents an important physiological parameter for the diagnosis and management of multiple brain disorders. The clinical need for CBF measurements is further complicated by the desire to have a non-invasive method with high temporal resolution that can measure CBF over a wide range of blood flows and in a wide range of patients. Numerous techniques are available to measure CBF. Nuclear medicine approaches, such as single positron emission computed tomography (SPECT) and positron emission tomography (PET) rely on radioisotopes which can be problematic in the pediatric population. In contrast, MRI-based methods are non-invasive and the CBF information can be obtained in conjunction with other MRI techniques (i.e. diffusion weighted imaging or spectroscopy) which allows for a combined longitudinal assessment of CBF, morphology, and metabolism, to provide a more complete understanding of the developing pathophysiological mechanisms.

Arterial spin labeling (ASL) perfusion imaging uses arterial blood water as an endogenous diffusible tracer where radiofrequency (RF) pulses magnetically label the moving spins in flowing blood without the use of a contrast agent. After a time delay allowing for the magnetically labeled blow to flow into the brain, "labeled" images are acquired. Separate control images are also acquired, without labeling and the difference between the two sets of imaged provides a measure of perfusion. Since gadolinium-based contrast agents are not required, the ASL perfusion technique is completely non-invasive. In addition, ASL techniques are insensitive to blood-brain barrier permeability changes, which can occur after strokes or with tumors.

Because gadolinium-based contrast is not used, the ASL technique has an inherently lower sensitivity than DSC-PWI. To date, there are a number of commercially available ASL techniques that differ in their labeling schemes, which has contributed to the difficulty in obtaining consistent results across different patient populations (pediatric, elderly, stroke, tumors). A number of recent reports using pseudo-continuous ASL (pCASL) have been published and show increased reliability across different patient populations. Moreover, a recent consensus statement published by the International Society of Magnetic Resonance in Medicine Perfusion Study Group recommends the use of pCASL labeling strategies for clinical applications.

The objectives of this study is to determine the accuracy and reliability of a newly developed pCASL sequence and post-processing software across multiple patient populations (neonate to elderly) and pathological processes.

ELIGIBILITY:
Inclusion Criteria:

* Any person between the ages of 18-90 years, who is undergoing routine magnetic resonance imaging (MRI) of the head with or without contrast at Loma Linda University Medical Center.
* Must be eligible for MRI (no electronic or metal implants that are not MR compatible).

Exclusion Criteria:

* Electronic or metal implant that is not MRI safe, pregnancy or claustrophobia.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-05; Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Bartnik Olson, PhD, Principal Investigator — Loma Linda University Medical Center

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magentic Resonance Imaging
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: any person between age of 18-90
Arm/Group | Magentic Resonance Imaging
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Regional Cerebral Blood Flow Values of the Brain Measured Using Pseudo-continuous Arterial Spin Labeling (pCASL) MRI.
Description: The relative cerebral blood flow (CBF) in frontal, parietal, occipital gray matter and white matter regions, basal ganglia, thalami, and cerebellum will be measured using region of interest analysis to determine institutional normative values for healthy subjects.
Time Frame: single encounter
Population: control
Measure: Mean (Standard Deviation); unit: ml/100g/min
Arm/Group | Magentic Resonance Imaging
Number analyzed (Participants) | 1
ml/100g/min | 35.4 (5.7)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Magentic Resonance Imaging
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT02767609/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2014-04-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT02767609/Prot_SAP_001.pdf